CLINICAL TRIAL: NCT04152564
Title: The Cardio-pulmonary and Analgesic Effects of Pre-peritoneal Infusion VS Epidural Infusion of Levo - Bupivacaine on Patients Undergoing Major Upper Abdominal Cancer Surgery
Brief Title: Cardio-pulmonary and Analgesic Effects of Pre-peritoneal VS Epidural Infusion of L-bupivacaine on Abd. Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Mohammed Farghaly Abd El hamid Ahmed, assisstant lecturer, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 440
Record Dates: First submitted 2019-10-16; First posted 2019-11-05 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Abdominal Cancer
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- levo-bupivacaine continuous epidural infusion [CEI]) (Active Comparator): The epidural catheter will be placed via a paramedian approach as close as possible to the surgical procedure via the inter-vertebral space (from T7 to T10) so that the affected dermatomes of the surgical wound would receive the benefits of bupivacaine infusion. Proper placement of the catheter was verified through an aspiration test and a test dose (2 ml) of lidocaine 2%. At the end of surgery, a 14 ml bolus of L-bupivacaine 0.125 will be administered through the catheter and then a continuous rate of .1 ml/kg/h infusion of L-bupivacaine 0.125 will be delivered.
  Interventions: Procedure: levo-bupivacaine infusion via Thoracic epidural catheter
- Levo-bupivacaine continuous preperitoneal infusion [CPI]), (Active Comparator): At the end of surgery and after the closure of the peritoneal layer, the preperitoneal catheter will be allocated above the peritoneum within the musculofascial layer and secured to the skin with an occlusive dressing. Thereafter, a 20 ml bolus of L-bupivacaine 0.25% will be administered through the catheter and then a continuous fixed-rate infusion of L-bupivacaine 0.25% will be delivered.
  Interventions: Procedure: levo-bupivacaine infusion via preperitoneal catheter

INTERVENTIONS:
Procedure: levo-bupivacaine infusion via Thoracic epidural catheter — The epidural catheter will be placed via a paramedian approach as close as possible to the surgical procedure via the inter-vertebral space (from T7 to T10) so that the affected dermatomes of the surgical wound would receive the benefits of bupivacaine infusion
  Other Names: TEA
  Arms: levo-bupivacaine continuous epidural infusion [CEI])
Procedure: levo-bupivacaine infusion via preperitoneal catheter — At the end of surgery and after the closure of the peritoneal layer, the catheter will be allocated above the peritoneum within the musculofascial layer and secured to the skin with an occlusive dressing
  Arms: Levo-bupivacaine continuous preperitoneal infusion [CPI]),

SUMMARY:
60 Patients will be randomly assigned using computer generated randomization program (http://www.randomizer.org) into two groups, First group (Control group ,Group of continous epidural infusion [CEI]), where patients will receive continuous epidural infusion of L-bupivacaine 0.125 % at a rate of .1 ml/kg/h during the first 48 hours after surgery. Second group (Group of continous preperitoneal infusion [CPI]), where patients will receive continuous pre-peritoneal wound infusion with L-bupivacaine 0.25% at 10 ml/h during the first 48 hours after surgery.

DETAILED DESCRIPTION:
All patients will receive IV morphine when needed for a period of 48 hours with a PCA device programmed to deliver 1 mg/dose with a 10-minute lockout time without background infusion.

CEI group The epidural catheter will be placed via a paramedian approach as close as possible to the surgical procedure via the inter-vertebral space (from T7 to T10) so that the affected dermatomes of the surgical wound would receive the benefits of bupivacaine infusion. Proper placement of the catheter was verified through an aspiration test and a test dose (2 ml) of lidocaine 2%. At the end of surgery, a 14 ml bolus of L-bupivacaine 0.125 will be administered through the catheter and then a continuous rate of .1 ml/kg/h infusion of L-bupivacaine 0.125 will be delivered.

CPI group At the end of surgery and after the closure of the peritoneal layer, the catheter will be allocated above the peritoneum within the musculofascial layer and secured to the skin with an occlusive dressing. Thereafter, a 20 ml bolus of L-bupivacaine 0.25% will be administered through the catheter and then a continuous fixed-rate infusion of L-bupivacaine 0.25% will be delivered.

Outcome Measures The primary outcome will be the pulmonary effects including

. Respiratory mechanics: Forced Vital Capacity (FVC) &Forced Expiratory Volume in one second (FEV1) will be assessed preoperatively and at 12h, 24h and 48 hours postoperatively.

The Secondary outcome of the study will include the following:

* Cardiac enzymes: Troponin I and plasma BNP levels will be measured preoperatively and postoperative day 1 and day 2.
* Intensity of pain at rest and during pain-provoking movements (deep breathing, coughing, mobilization) measured by VAS pain score immediately postoperative then at 2, 4 ,6 ,12, 24 ,36 &48 hours after surgery.
* Hemodynamic variables including (systolic and diastolic BP, heart rate, oxygen saturation & respiratory rate) measured preoperatively (baseline measurement) then immediately postoperative and at 2, 4 ,6 ,12, 24 ,36 &48 hours after surgery.
* Blood gases will be drawn preoperatively and at 12 hour interval in the PACU for assessment of Oxygen tension (PO2) & Co2 tension (PCO2).

  * Morphine titration and dosage required in the post-anesthesia care unit (PACU).
  * IV PCA Total morphine consumption during first 48 hours postoperatively.
* Time of return of intestinal sounds.
* CVP will be measured preoperatively and at post anaesthesia care unit for crude assessment of cardiac function

  * Quality of night sleep assessed at 8:00 am on postoperative days 1 and 2 using a verbal numerical scale (VNS) ranging from 0 (poor quality) to 10 (excellent quality).
  * Patient satisfaction with the quality of postoperative analgesia 48 hours after the end of surgery, assessed on a 5-point scale (completely dissatisfied, dissatisfied, not satisfied nor dissatisified, satisfied or completely satisfied [34].
  * side effects, including hemodynamic variables (hypotension & bradycardia), supine hypotension ,shivering ,bladder distension and PONV.
* Complications of Thoracic epidural as (Inadvertent intrathecal injection, Spinal hematoma, Spinal abscess, superficial cellulites, PDPH, Nerve injury &Back pain) will be assessed and managed

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected to major upper abdominal cancer surgery.
* The enrolled age will be from 18 years to 70 years
* ASA, I-III and NYHA, I-III.

Exclusion Criteria:

* ASA physical status and NYHA >III,
* pregnant women,
* body mass index >40 kg/m2,
* preoperative opioid consumption,
* Contraindications or patient's refusal of epidural analgesia, and inability to use a PCA device.
* Contraindications of use of spirometry device :

A) Cerebral aneurysm, Recent brain surgery, recent concussion, recent eye surgery& Significant glaucoma.

B) Recent sinus surgery or middle ear surgery or infection. C) Pneumothorax, Significant aortic aneurysm, Recent thoracic surgery or Recent abdominal surgery .

D) Systemic hypotension or severe hypertension (eg, >200/120 mmHg), Significant atrial/ ventricular arrhythmia , Noncompensated heart failure , Recent myocardial infarction or pulmonary embolus.

E) History of syncope related to forced exhalation/cough. F) Active tuberculosis , Hemoptysis or oral bleeding . 7-Uncooperative patients regarding use of spirometry [Inability to follow directions (eg, confusion, dementia, young age, language barrier)].

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
change in Respiratory mechanics | preoperative-Day 1 & Day2 postoperative
  Forced Vital Capacity (FVC) &Forced Expiratory Volume in one second (FEV1) will be assessed preoperativly and at Day 1 & Day2 postoperative.

SECONDARY OUTCOMES:
change in Cardiac enzymes levels | preoperatively and postoperative Day 1 and Day 2.
  Troponin I and plasma BNP levels will be measured preoperatively and postoperative day 1 and day 2.
change in Visual analogue pain score | immediately postoperative then at 2 hours, 4hours ,6hours ,12hours, 24hours ,36hours &48 hours after surgery
  Intensity of pain at rest and during pain-provoking movements (deep breathing, coughing, mobilization) measured by VAS pain score with 11points where 0 means no pain,10 means sever pain

OTHER OUTCOMES:
Morphine titration and dosage required in the post-anesthesia care unit (PACU). | first 48 hours postoperatively.
  IV PCA Total morphine consumption during first 48 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: samy AA erfan, professor, Study Director — dean of SECI
Locations (1):
- South Egypt Cancer Inistitute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No